CLINICAL TRIAL: NCT00393978
Title: Quetiapine Plus Topiramate or Placebo for Bipolar Mania & Cannabis Use in Adolescents
Brief Title: Efficacy Study of Quetiapine Plus Topiramate for Reducing Cannabis Consumption and Bipolar Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Melissa Delbello, Professor, University of Cincinnati
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA; R01DA022221 (NIH)
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Results first posted 2017-08-29 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2016-05

CONDITIONS: Bipolar Disorder; Cannabis-Related Disorder
Keywords: Bipolar mania; Cannabis consumption
MeSH Terms: conditions — Bipolar Disorder; Marijuana Abuse | interventions — Quetiapine Fumarate; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine and Placebo (Placebo Comparator): Quetiapine and Placebo
  Interventions: Drug: Quetiapine and placebo
- Quetiapine and Topiramate (Active Comparator): Quetiapine and Topiramate
  Interventions: Drug: Quetiapine and Topiramate

INTERVENTIONS:
Drug: Quetiapine and placebo — placebo (titrated to 150-300 mg/day) in combination with quetiapine (titrated to 400-800 mg/day).
  Other Names: quetiapine
  Arms: Quetiapine and Placebo
Drug: Quetiapine and Topiramate — topiramate (titrated to 150-300 mg/day) in combination with Quetiapine (titrated to 400-800 mg/day).
  Arms: Quetiapine and Topiramate

SUMMARY:
The objectives of this study are to determine whether this treatment may be useful for reducing cannabis consumption; reducing symptoms of bipolar mania; and weight mitigation therapy for individuals on psychopharmacotherapy.

DETAILED DESCRIPTION:
The purpose of this research study is to study the effects (both good and bad) of combining medicines, called quetiapine and topiramate, for treating your symptoms, and other children and adolescents' symptoms, of bipolar mania (an illness with periods of elation, excessive excitement, irritability, high energy, racing thoughts, poor sleep, poor judgment, reckless behavior). It is estimated that 1% of the population of adolescents in the United States has bipolar disorder. The purpose of this research study is also to study the effects (both good and bad) of combining the same two medicines, quetiapine and topiramate, for reducing your use, and other children and adolescents' use, of cannabis (commonly referred to as "pot"). It is estimated that 30.5% of adolescents in the United States have used cannabis at least once in their lifetime. Additionally, the purpose of this research is to look at how bipolar disorder and cannabis use effects brain chemicals and function.

Quetiapine (marketed under the brand name Seroquel) has been approved by the FDA since 1997 to help adults who suffer from schizophrenia (an illness of feeling, thought, perception and behavior). On January 12, 2004, the FDA approved quetiapine for the treatment of bipolar symptoms in adults. As of December 2009, Quetiapine has now been approved by the FDA for use in adolescents (13-17 years of age) for the treatment of schizophrenia and for the treatment of manic episodes associated with bipolar I disorder in children and adolescents (10-17 years of age). Bipolar disorder is an illness characterized by recurrent mood swings including mania (i.e., periods of elation, excessive excitement, irritability, high energy, racing thoughts, poor sleep, poor judgment, reckless behavior) and clinical depression (i.e., a depressed mood, loss of interest in activities and disruption of sleep, appetite and energy). This study is being carried out to see if quetiapine is effective and safe for treatment of children and adolescents who have the symptoms of bipolar mania. This study is also being carried out to see if quetiapine, in combination with topiramate, will further reduce bipolar mania and reduce cannabis use.

As of December 2, 2009, the US Food and Drug Administration (FDA) approved SEROQUEL (quetiapine fumarate) tablets for the treatment of schizophrenia in adolescents (13-17 years of age) as monotherapy, and for the acute treatment of manic episodes associated with bipolar I disorder in children and adolescents (10-17 years of age), both as monotherapy and as an adjunct to lithium or divalproex.

Topiramate (marketed under the brand name Topamax) is approved by the U.S. FDA for the prevention of migraine headaches in adults. The FDA has also approved topiramate for epilepsy (a seizure disorder) and for use as adjunctive therapy (meaning in combination with other medicines) for partial onset seizures in adults. Topiramate is not approved by the FDA for use in adults or for use in children and adolescents who have bipolar disorder. This study is being done to see if topiramate, in combination with quetiapine, will reduce bipolar mania and reduce cannabis use.

The FDA has declared research studies with MRI field strengths up to and including 8 Tesla (a measure of field strength) as non-significant risk. This research study uses an MRI with a field strength of 4 Tesla.

ELIGIBILITY:
Inclusion/Exclusion Criteria Inclusion Criteria: To be included, all subjects must…

* have an authorized parent/legal guardian who understands the nature of the study and who provides written informed consent if the study subject is younger than 18 years of age. Additionally, each subject must provide assent to the study;
* be fluent in English;
* be 12 to 21 years of age, inclusive;
* be using a medically accepted means of contraception (i.e., oral contraceptives and barrier methods (diaphragm or condom), medroxyprogesterone acetate injectable suspension, abstinence) if female and of menarche. Oral contraceptives alone are not acceptable means of contraception because concomitant use of topiramate and low estrogen oral contraceptive pills may lead to oral contraceptive failure;
* have a diagnosis of bipolar I disorder in a current manic or mixed episode, in addition to a cannabis use disorder (which includes abuse or dependence) within 28 days prior to screening, as determined by the WASH-U-KSADS;
* have an initial YMRS total score of >16 at screening and baselines;
* use cannabis a minimum of twice per week on average during the 28 days prior to screening.

Exclusion Criteria: Subjects will not be eligible for participation if they…

* have a known history of mental retardation;
* are acutely intoxicated, and thus impaired;
* have manic or depressive symptoms resulting entirely from acute medical illness or acute intoxication or withdrawal from drugs or alcohol, as determined by medical evaluation and rapid symptom resolution;
* have clinically significant alcohol or other drug withdrawal symptoms, as determined by vital signs, The Clinical Institute Withdrawal Assessment for Alcohol Scale - Revised (CIWA-Ar)24, and physician interview;
* have any unstable medical or neurological illness as determined by a study physician;
* have laboratory abnormalities >3 times upper limits of established normal values;
* as females, have a positive serum (screening and week 16) or urine pregnancy test (at baseline and weeks 1-16), are lactating, or are not practicing a reliable form of birth control;
* have a history of nephrolithiasis, since topiramate has been associated with an elevated risk of kidney stones;
* require concurrent treatment with mood stabilizers, anticonvulsants, or antidepressants
* require concurrent treatment with carbonic anhydrase inhibitors.
* have significant suicidal ideation
* have been treated for a substance use disorder during 28 days prior to screening or are court-ordered to treatment for substance use to ensure that, if we detect a change in use with topiramate treatment, it is likely not due to these other confounding factors that might influence substance use. Peer support groups are not considered treatment for substance use. **Patients can be enrolled into the study that are already enrolled in a court ordered substance treatment, for at least 1 month prior to study enrollment, if they still meet the minimum cannabis use criterion.**
* have been diagnosed or treated for an eating disorder, to make sure any weight loss does not contribute to an already underlying condition
* have a family history of glaucoma, since topiramate has been associated with an elevated risk of glaucoma;
* have a history of non-response or hypersensitivity to quetiapine or topiramate;
* if scanning, have claustrophobia and/or contraindicated for magnetic resonance scanning (i.e. intraocular metallic objects, braces, cochlear implants, pacemakers, or other electrical, mechanical, or magnetically activated implants); and
* if scanning, have a history of significant head trauma (i.e. injury resulting in loss of consciousness for greater than five minutes).

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa P DelBello, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farrow JE, DelBello MP, Patino LR, Blom TJ, Welge JA. A Double-Blind, Placebo-Controlled Study of Adjunctive Topiramate in Adolescents With Co-Occurring Bipolar and Cannabis Use Disorders. JAACAP Open. 2024 Sep 7;2(4):290-300. doi: 10.1016/j.jaacop.2024.08.002. eCollection 2024 Dec. PMID 39697396

RESULTS

PARTICIPANT FLOW:
Groups:
- Quitiapine + Placebo: Quetiapine + Placebo
  quetiapine + placebo: placebo (titrated to 150-300 mg/day) in combination with quetiapine (titrated to 400-800 mg/day).
- Quetiapine + Topiramate: Quetiapine + Topiramate
  Quetiapine + Topiramate: topiramate (titrated to 150-300 mg/day) in combination with Quetiapine (titrated to 400-800 mg/day).
Period: Overall Study
Arm/Group | Quitiapine + Placebo | Quetiapine + Topiramate
Started | 37 | 38
Completed | 21 | 18
Not Completed | 16 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quitiapine + Placebo | Quetiapine + Topiramate | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 38 | 75
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.1 (2.1) | 17.7 (2.1) | 17.4 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 19 | 18 | 37
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change in Joints Per Week
Description: Change in timeline follow-back self-reported of joint equivalents per week from baseline to 16 weeks.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: joints
Groups:
- Quitiapine and Placebo: Quetiapine and Placebo
  Quetiapine and placebo: placebo (titrated to 150-300 mg/day) in combination with quetiapine (titrated to 400-800 mg/day).
Arm/Group | Quitiapine and Placebo | Quetiapine and Topiramate
Number analyzed (Participants) | 37 | 38
joints | -10.1 (27.2) | -10.7 (18.4)

2. Primary Outcome: Change in Percent Days of Cannabis Use Per Week
Description: Change in percent days of cannabis use per week from baseline to week 16.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: cannabis use
Arm/Group | Quitiapine and Placebo | Quetiapine and Topiramate
Number analyzed (Participants) | 37 | 38
cannabis use | -29.9 (41.1) | -43.5 (38.1)

ADVERSE EVENTS:
Time Frame: Over a period of 3 years
Arm/Group | Quitiapine + Placebo | Quetiapine + Topiramate
Serious Adverse Events (participants affected / at risk) | 6/37 | 5/38
Other Adverse Events (participants affected / at risk) | 30/37 | 23/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quitiapine + Placebo (N=37) | Quetiapine + Topiramate (N=38)
Pregnancy (Reproductive system and breast disorders) | 1 | 0
Hospitalization (Psychiatric disorders) | 5 | 4 — Exacerbation of illness
Increased Suicidal Ideation (Psychiatric disorders) | 0 | 1 — Increased suicidal ideation during hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quitiapine + Placebo (N=37) | Quetiapine + Topiramate (N=38)
Difficulty falling asleep (General disorders) | 20 | 12
Difficulty staying asleep (General disorders) | 20 | 12
Excitement (General disorders) | 0 | 5
Dry Mouth (General disorders) | 30 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No